CLINICAL TRIAL: NCT00374972
Title: Combined Hormonal Versus Progestin Only Contraception During Lactation
Status: Withdrawn | Type: Observational
Why Stopped: difficulty in recruitment. lack of sponsorship
Sponsor: Shaare Zedek Medical Center (Other)
Collaborators: Organon (Industry)
Other Study IDs: 40106
Record Dates: First submitted 2006-09-11; First posted 2006-09-12 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-04

CONDITIONS: Lactation
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (2):
- combined contraceptives: combined contraceptives
- pregesterone only contraceptives: pregesterone only contraceptives

SUMMARY:
Objective: To determine and compare the effect of low dose estrogen combined hormonal contraceptives and progestin-only contraceptives on lactation.

The subjects will be drawn from a healthy obstetric population in each center, where possible preliminary contact during antenatal period. At the postpartum visit, subjects that express their wish for a hormonal contraceptive method will be offered enrollment. After obtaining an informed consent the participants will be allocated according to their free wish to either receive a combined preparation containing 0.02 mg ethylestradiol and 0.15 mg desogestrel (Mercilon, Organon) or a progestin only pill containing 0.075 mg desogestrel (Cerazette, Organon). Demographic, habits and perinatal data will be collected and stored to analysis.

Frequency and methods of observation: All women will be followed at 6 (baseline), 9 and 12 weeks post - partum. Instruction will be given as to recording information on intercurrent disease, frequency of nursing and use of complementary formula supplements. Maternal BMI calculation ( weight/height2) will be obtained at first visit.

The objective is to compare the capacity of the breast to secrete milk under standard conditions and evaluate the influence of different hormonal contraception means. Thus samples will be collected at 6 weeks (enrollment) and the 9 and 12 weeks visits. An Egnell pump will be used for a maximum of 20 minutes form from both breasts, simulating a regular breast feeding. A total of 10 ml aliquot will be taken for composition analysis and the rest will be offered to the infant. The milk volume/feeding will be estimated and expressed in ml/feeding and multiplied by the number of feedings reported.

Outcome variables: Milk volume, infant growth at each visit and biochemical markers of milk analysis : lipid, casein and carbohydrate content

ELIGIBILITY:
Inclusion Criteria:

* healthy

Exclusion Criteria:

* mothers to infants that their weight will be below the 10th percentile
* mothers to infants sensitive to milk

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2006-06 (Actual); Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naama Srebnik, MD, Principal Investigator — A resident at the Shaare Zedek Medical Center; Surina Grisaru-Granovsky, Study Director — A senior doctor at the Shaare Zedek Medical Center